CLINICAL TRIAL: NCT01140802
Title: A Study of the Gut Microbiota in the Healthy Population, Patients With Inflammatory Bowel Disease and Their Relatives (IBD Microbe Study
Brief Title: Gut Microbiota in the Healthy Population, Inflammatory Bowel Disease Patients, and Their Relatives
Status: Terminated | Type: Observational
Why Stopped: Due to study plan
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: IBD Microbe
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Inflammatory Bowel Disease
Keywords: First degree relatives; Crohn's disease; Ulcerative colitis; Healthy control
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum DNA will be collected and stored only if patients have provided consent separately. All serum DNA blood samples will be anonymised. Genetic results will not be made available to individual patients in a future date as there is no evidence to support genetic testing for risk prediction in routine practice, but these large scale genetic results will be useful to identify relevant future therapeutic targets for treatment of IBD. 10 ml of blood will be collected in EDTA tubes and stored at minus 80 degrees C, These samples will be transported to China for analysis at a later date.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- IBD patients: Crohn's disease or ulcerative colitis patients
- Healthy controls (non-IBD): Patients comprise ethnicity - matched patients undergoing colonoscopy for polyp or colorectal cancer screening, or rectal bleeding
- Relatives of IBD patients: They will be a first degree relative of a IBD patient.

SUMMARY:
The aim of this study is to compare the gut microbiota in Chinese patients with Inflammatory Bowel Disease (IBD) in Hong Kong with that of healthy controls, compare the gut microbiota in IBD patients in a developing country (low but increasing IBD incidence, Hong Kong) with those in a developed country (high incidence, Australia), compare the gut microbiota in Chinese patients with IBD in Hong Kong with the microbiota of their non-IBD affected parents and siblings.

DETAILED DESCRIPTION:
Crohn's disease and ulcerative colitis are chronic inflammatory disorders of the gut that cause major life-long disability. Afflicting mostly young people at an age when they are most active both in their private and professional life, inflammatory bowel disease (IBD) represents an important public health problem affecting both the patients education, working abilities, social life and quality of life. Previously a disease predominantly of the West, there is now a marked increase in the incidence of IBD in Hong Kong. The cause of this dramatic increase over the last decade is unknown. Genetic factors, environmental factors and the gut bacteria may play a role in disease development. This study aims to explore the factors that may be contributing to, or causing, the rise of IBD in Hong Kong. The investigators propose to study the gut bacteria in Chinese patients with IBD compared with non-IBD patients, and healthy relatives of IBD patients. IBD patients will be prospectively recruited, blood samples will be obtained for serology and genotyping, stool samples and biopsies will be collected during routine colonoscopy for microbiota analysis. Bloods, stool and tissue gut microbiota from non-IBD patients will be collected for comparison. Studying gut microbiota, genetics and environmental factors in populations with changing incidence of IBD offers the greatest hope of identifying potentially important causative factors for disease.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥18 with a diagnosis of Crohn's disease or ulcerative colitis defined by endoscopy, radiology and histology, patients on stable medication and informed consent obtained

Control group:

Healthy controls (non-IBD patients) will comprise ethnicity - matched patients undergoing colonoscopy for polyp or colorectal cancer screening, or rectal bleeding. Controls will be excluded if they have previously been diagnosed with IBD or if they have a first or second degree relative with IBD.

Relatives group:

Relatives of patients will be aged between 16 and 35 years. They will be a first degree relative of a patient. Relatives older than 35 will not be recruited to maximise the chance of including some individuals who will develop IBD in the future. Relatives will be contacted either via the patient or directly by telephone by the investigators. They will be invited to attend for a screening meeting to assess eligibility and to receive the information sheets. They will undergo a flexible sigmoidoscopy/colonoscopy for biopsies once fully consented.

Exclusion Criteria:

* Patient group:

  1. current infection with an enteric pathogen,
  2. use of antibiotics within the last month,
  3. consumption of any probiotic or prebiotic within the last month,
  4. imminent need for surgery,
  5. requiring hospitalization,
  6. pregnancy or lactation,
  7. short bowel syndrome
  8. previous proctocolectomy
  9. significant hepatic, renal, endocrine, respiratory, neurological or cardiovascular disease as determined by the principal investigator,
  10. if they have a history of cancer with a disease free state of less than two years

Control and Relative group:

1. previously been diagnosed with IBD
2. they have a first or second degree relative with IBD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Crohn's disease or ulcerative colitis patients as the case groups, Patients attend clinics or endoscopy for functional upper gastrointestinal diseases or screening colonoscopy as the control group, and the first degree relatives of IBD patients as the relative group
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To identify specific gut microbiota in IBD patients | 2 years
  Dominant species from colonic tissue and stool samples including bacteroides, bifidobacteria, firmucutes (using microarray analysis and pyrosequencing)

SECONDARY OUTCOMES:
To identify environmental risk factors | 2 years
  A validated Enviromental risk factor questionnaire by International Organisation of Inflammatory Bowel Disease
To identify genetic differences among IBD patients, their relatives and the control subjects | 2 years
  To measure common known genetic variants including NOD2 mutation, IL23R, TNFSF15, etc from blood samples
To identify disease characteristics among IBD patients | 2 years
  Disease characteristics including disease behavior, disease location and progression according to Montreal Classification.

CONTACTS AND LOCATIONS:
Overall Officials: Siew C NG, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No